CLINICAL TRIAL: NCT00908271
Title: Study of the Absolute Oral Bioavailability of Dapagliflozin in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: MB102-059
Record Dates: First submitted 2009-05-22; First posted 2009-05-25 (Estimated); Last update posted 2016-10-17 (Estimated); Status verified 2016-10

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — dapagliflozin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Dapagliflozin (Other): PO and IV
  Interventions: Drug: Dapagliflozin

INTERVENTIONS:
Drug: Dapagliflozin — Tablet and IV solution, Oral and IV, 10 mg po and 100 µg IV, Single oral dose followed by a single IV dose (IV dose administered at 1h after oral dose), 1 day

SUMMARY:
The purpose of this study is to estimate the absolute oral bioavailability of dapagliflozin.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects (ages 18 to 45) as determined by medical history, physical examination, 12-lead electrocardiogram (ECG), and clinical laboratory evaluations will be eligible to participate in the study

Exclusion Criteria:

* Evidence of organ dysfunction or any clinically significant deviation from normal in physical examination, vital signs, ECG or clinical laboratory determinations
* Participation in a radiolabeled investigational study drug trial within 12 months prior to admission to the clinical facility
* Exposure to significant radiation within 12 months prior to admission to the clinical facility

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 7 (Actual)
Dates: Start 2009-07; Primary Completion 2009-08 (Actual); Study Completion 2009-08 (Actual)

PRIMARY OUTCOMES:
Absolute oral bioavailability | Within the 3 days after study drug administration

SECONDARY OUTCOMES:
Adverse events (AE) | Within the 3 days after study drug administration
Vital signs | Within the 3 days after study drug administration
Clinical safety labs | Within the 3 days after study drug administration
Electrocardiograms (ECGs) | Within the 3 days after study drug administration

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- Covance Clinical Research Unit, Inc., Madison, Wisconsin, United States

REFERENCES:
- See also: MB102-059_redacted _CSR _synopsis — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_MED_7111&studyid=3649&filename=MB102-059_redacted%20_CSR%20_synopsis.pdf